CLINICAL TRIAL: NCT02870855
Title: Effect of Intrauterine Injection of Human Chorionic Gonadotropin Before Embryo Transfer on Clinical Pregnancy Outcome in Repeated Implantation Failure Patients
Brief Title: Effect of Intrauterine Injection of HCG on Pregnancy Outcome in Repeated Implantation Failure Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Entry criteria were changed, investigator have registrated a new trials.
Sponsor: Reproductive & Genetic Hospital of CITIC-Xiangya (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KYXM-201604
Record Dates: First submitted 2016-08-14; First posted 2016-08-17 (Estimated); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HCG group (Experimental): intrauterine injection of HCG before blastocyst transfer
  Interventions: Drug: intrauterine injection of HCG
- Control group (No Intervention): blastocyst transfer

INTERVENTIONS:
Drug: intrauterine injection of HCG — intrauterine injection of HCG berore blastocyst transfer
  Arms: HCG group

SUMMARY:
Repeated implantation failure（RIF） is a insurmountable bottleneck in assisted reproductive technology, many studies have considered that the cause of two-thirds of implant failure is the decreased endometrial receptivity. Human chorionic gonadotropin (hCG) is an early pre-plant signal molecule secreted by the embryo, it can promote endometrial proliferation, increase blood flow and promote embryonic adhesion and inhibit self-regulate apoptosis of trophoblast cells. Previous studies showed that: intrauterine injection of HCG before embryo transfer can improve clinical outcomes in IVF/Intracytoplasmic sperm injection(ICSI). But some studies found that the intrauterine injection of HCG can not significantly improve the success rate of blastocyst transfer, and the reason may be the intrauterine injection of HCG time is too late to significantly increase the implantation rate. Would ahead of intrauterine injection of HCG be more effective? Thus, the patients of repeated implantation frozen embryo cycle according to the random principle accepted two kinds of transplants ways: ①intrauterine injection of HCG before blastocyst transfer; ②blastocyst transfer. Try to understand whether intrauterine injection of HCG can significantly improve the clinical pregnancy rate of blastocyst transfer in repeated implantation failure patients.

ELIGIBILITY:
Inclusion Criteria:

* women with unexplained RIF(two to four previous embryo transfers without achieving pregnancy);
* age<36 years;
* frozen embryo transfer cycles

Exclusion Criteria:

* polycystic ovary syndrome
* uterine abnormalities (double uterus, bicornuate uterus, unicornuate uterus and uterine mediastinum)
* intrauterine adhesions
* endometriosis
* adenomyosis
* hydrosalpinx
* uterine fibroids (submucosal fibroids, non-mucosal fibroids > 4 cm and / or endometrial pressure)
* thydroid dysfunction and hyperprolactinemia

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2017-07-28 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2018-01-01 (Actual)

PRIMARY OUTCOMES:
clinical pregnancy rate | Until 28 day after embryo transferred
  clinical pregnancy rate

SECONDARY OUTCOMES:
spontaneous abortion rate | until 28 day after embryo transferred
  spontaneous abortion rate
ectopic pregnancy rate | until 28 day after embryo transferred
  ectopic pregnancy rate

CONTACTS AND LOCATIONS:
Locations (1):
- Reproductive & Genetic Hospital of CITIC-XIANGYA, Changsha, Hunan, China